CLINICAL TRIAL: NCT01459965
Title: Endoscopic Palliation of Malignant Biliary Tract Obstruction: Emphasis on Improvement in Quality of Life
Brief Title: Stenting Malignant Jaundice for Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: American Society for Gastrointestinal Endoscopy (Other); American College of Gastroenterology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 9307-04
Record Dates: First submitted 2011-10-21; First posted 2011-10-26 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Bile Duct Neoplasms Malignant
Keywords: Jaundice; Biliary stents; Palliation; Quality of Life; Endoscopic Retrograde Cholangiography
MeSH Terms: conditions — Jaundice | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10 French Stent (Active Comparator): 10 French biliary plastic stent
  Interventions: Procedure: ERCP with 10 French biliary plastic stent placement
- 11.5 French stent (Active Comparator): 11.5 French biliary plastic stent
  Interventions: Procedure: ERCP with 11.5 French biliary plastic stent

INTERVENTIONS:
Procedure: ERCP with 10 French biliary plastic stent placement — Stent placement of a 10 French biliary plastic stent
  Arms: 10 French Stent
Procedure: ERCP with 11.5 French biliary plastic stent — biliary plastic stent placement
  Arms: 11.5 French stent

SUMMARY:
Endoscopic stent insertion is considered the method of choice for palliation of malignant bile duct obstruction (MBDO). However, it can cause complications and requires periodic stent exchanges. While endoscopic stenting is clearly indicated for relief of cholangitis or refractory pruritus, its role in patients with jaundice alone is less clear. Endoscopic stenting for this relative indication might be justified, if there is a significant improvement in quality of life (QOL) of such patients. The aim of the investigators study was to determine whether endoscopic stenting for MBDO results in improved QOL.

DETAILED DESCRIPTION:
Most malignant tumors causing bile duct obstruction, such as pancreatic adenocarcinoma, gallbladder carcinoma or cholangiocarcinoma, have an extremely poor prognosis. At the time of diagnosis the majority of these tumors will be unresectable with a median survival of 4-6 months. Palliation is the goal for those patients with unresectable tumors and limited survival and for those at high risk for attempts at curative resection.

Endoscopic retrograde cholangiopancreatography (ERCP) with endoscopic stent insertion is considered the method of choice for palliative treatment of malignant bile duct obstruction (MBDO). However, it can cause complications, such as pancreatitis, bleeding, perforation, cholangitis and stent migration in a significant proportion of treated patients. Clogging of plastic stents is a predictable consequence and requires periodic stent exchanges with attendant risks and costs. While endoscopic stenting is clearly indicated for relief of cholangitis or refractory pruritus, the role of stenting in patients with jaundice alone, abdominal pain, or failure to thrive due to malignancy is less clear. Given the risk for complications and costs, endoscopic therapy might be justified in these clinical scenarios if quality of life (QOL) is significantly improved. A few available studies have demonstrated improved QOL in stented patients. However, these studies include a small number of patients and/or are retrospective in design. Therefore, more evidence to support routine palliative biliary drainage in patients with MBDO is desired.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected or proven malignant biliary obstruction who were unresectable or inoperable and were undergoing ERCP and biliary stenting for biliary depression.

Exclusion Criteria:

* Had previously undergone biliary stenting
* Surgery was planned
* A guidewire could not be passed through the stricture
* Suspected survival of < 3 months
* Impending duodenal obstruction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 1993-07; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Documented change in Quality Of Life | 180 days after stent insertion
  Documented change in QOL over the first month and over six months after successful biliary drainage compared with that before the procedure. The FACT-G questionnaire administered at baseline, at 1 month after stent insertion and at 180 days after stent insertion was used to assess this outcome. Change from baseline was analyzed at each of these time points separately.

SECONDARY OUTCOMES:
Documented change in symptoms and concerns specific for patients with MBDO | 180 days after stent placement
  An additional 10 item questionnaire was administered at baseline, at 1 month after biliary stenting and at 180 days after biliary stenting.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Sherman, MD, Principal Investigator — Indiana University School of Medicine; Glen A Lehman, MD, Principal Investigator — Indiana Univesity Medical Center; James Frankes, MD, Principal Investigator — Rockford GE Associates; John Johanson, MD, Principal Investigator — Rockford GE Associates; Tahir Qaseem, MD, Principal Investigator — MaineHealth; Douglas Howell, MD, Principal Investigator — MaineHealth

REFERENCES:
- [Background] Jemal A, Thomas A, Murray T, Thun M. Cancer statistics, 2002. CA Cancer J Clin. 2002 Jan-Feb;52(1):23-47. doi: 10.3322/canjclin.52.1.23. PMID 11814064
- [Background] Lowy AM. From bad to worse: prognostic factors in pancreatic cancer. Ann Surg Oncol. 2004 Feb;11(2):117-8. doi: 10.1245/aso.2004.12.930. No abstract available. PMID 14761910
- [Background] Lowenfels AB, Maisonneuve P, Boyle P (1998) Epidemiology of pancreatic cancer. In: Howard J, Idezuki Y, Ihse I, Prinz R, eds. Surgical Diseases of the Pancreas. 3rd ed. Baltimore: Williams & Wilkins, 433-439
- [Background] Speer AG, Cotton PB, Russell RC, Mason RR, Hatfield AR, Leung JW, MacRae KD, Houghton J, Lennon CA. Randomised trial of endoscopic versus percutaneous stent insertion in malignant obstructive jaundice. Lancet. 1987 Jul 11;2(8550):57-62. doi: 10.1016/s0140-6736(87)92733-4. PMID 2439854
- [Background] Andersen JR, Sorensen SM, Kruse A, Rokkjaer M, Matzen P. Randomised trial of endoscopic endoprosthesis versus operative bypass in malignant obstructive jaundice. Gut. 1989 Aug;30(8):1132-5. doi: 10.1136/gut.30.8.1132. PMID 2475392
- [Background] Motte S, Deviere J, Dumonceau JM, Serruys E, Thys JP, Cremer M. Risk factors for septicemia following endoscopic biliary stenting. Gastroenterology. 1991 Nov;101(5):1374-81. doi: 10.1016/0016-5085(91)90091-x. PMID 1936809
- [Background] Tarnasky PR, Cunningham JT, Hawes RH, Hoffman BJ, Uflacker R, Vujic I, Cotton PB. Transpapillary stenting of proximal biliary strictures: does biliary sphincterotomy reduce the risk of postprocedure pancreatitis? Gastrointest Endosc. 1997 Jan;45(1):46-51. doi: 10.1016/s0016-5107(97)70301-8. PMID 9013169
- [Background] Margulies C, Siqueira ES, Silverman WB, Lin XS, Martin JA, Rabinovitz M, Slivka A. The effect of endoscopic sphincterotomy on acute and chronic complications of biliary endoprostheses. Gastrointest Endosc. 1999 Jun;49(6):716-9. doi: 10.1016/s0016-5107(99)70288-9. PMID 10343215
- [Background] Giorgio PD, Luca LD. Comparison of treatment outcomes between biliary plastic stent placements with and without endoscopic sphincterotomy for inoperable malignant common bile duct obstruction. World J Gastroenterol. 2004 Apr 15;10(8):1212-4. doi: 10.3748/wjg.v10.i8.1212. PMID 15069728
- [Background] Johanson JF, Schmalz MJ, Geenen JE. Incidence and risk factors for biliary and pancreatic stent migration. Gastrointest Endosc. 1992 May-Jun;38(3):341-6. doi: 10.1016/s0016-5107(92)70429-5. PMID 1607087
- [Background] Speer AG, Cotton PB, Rode J, Seddon AM, Neal CR, Holton J, Costerton JW. Biliary stent blockage with bacterial biofilm. A light and electron microscopy study. Ann Intern Med. 1988 Apr;108(4):546-53. doi: 10.7326/0003-4819-108-4-546. PMID 2450501
- [Background] Frakes JT, Johanson JF, Stake JJ. Optimal timing for stent replacement in malignant biliary tract obstruction. Gastrointest Endosc. 1993 Mar-Apr;39(2):164-7. doi: 10.1016/s0016-5107(93)70058-9. PMID 8388345
- [Background] Ballinger AB, McHugh M, Catnach SM, Alstead EM, Clark ML. Symptom relief and quality of life after stenting for malignant bile duct obstruction. Gut. 1994 Apr;35(4):467-70. doi: 10.1136/gut.35.4.467. PMID 7513672
- [Background] Pereira-Lima JC, Jakobs R, Maier M, Kohler B, Benz C, Martin WR, Riemann JF. Endoscopic stenting in obstructive jaundice due to liver metastases: does it have a benefit for the patient? Hepatogastroenterology. 1996 Jul-Aug;43(10):944-8. PMID 8884318
- [Background] Luman W, Cull A, Palmer KR. Quality of life in patients stented for malignant biliary obstructions. Eur J Gastroenterol Hepatol. 1997 May;9(5):481-4. doi: 10.1097/00042737-199705000-00013. PMID 9187881
- [Background] Abraham NS, Barkun JS, Barkun AN. Palliation of malignant biliary obstruction: a prospective trial examining impact on quality of life. Gastrointest Endosc. 2002 Dec;56(6):835-41. doi: 10.1067/mge.2002.129868. PMID 12447294
- [Background] Wagh MS, de Bellis M, Fogel EL, Frakes JT, Johanson JF, Qaseem T, Howell DA, Lehman GA, Sherman S. Multicenter Randomized Trial of 10-French versus 11.5-French Plastic Stents for Malignant Biliary Obstruction. Diagn Ther Endosc. 2013;2013:891915. doi: 10.1155/2013/891915. Epub 2013 May 2. PMID 23737656
- [Background] Cella DF, Tulsky DS, Gray G, Sarafian B, Linn E, Bonomi A, Silberman M, Yellen SB, Winicour P, Brannon J, et al. The Functional Assessment of Cancer Therapy scale: development and validation of the general measure. J Clin Oncol. 1993 Mar;11(3):570-9. doi: 10.1200/JCO.1993.11.3.570. PMID 8445433
- [Background] Cheung YB, Goh C, Thumboo J, Khoo KS, Wee J. Variability and sample size requirements of quality-of-life measures: a randomized study of three major questionnaires. J Clin Oncol. 2005 Aug 1;23(22):4936-44. doi: 10.1200/JCO.2005.07.141. PMID 16051946
- [Background] Steel JL, Eton DT, Cella D, Olek MC, Carr BI. Clinically meaningful changes in health-related quality of life in patients diagnosed with hepatobiliary carcinoma. Ann Oncol. 2006 Feb;17(2):304-12. doi: 10.1093/annonc/mdj072. Epub 2005 Dec 15. PMID 16357021
- [Background] Hahn EA, Cella D, (1997) Unbiased quality of life measurement across literacy levels and mode of administration. Qual Life Res 6:654.
- [Background] Yost KJ, Sorensen MV, Hahn EA, Glendenning GA, Gnanasakthy A, Cella D. Using multiple anchor- and distribution-based estimates to evaluate clinically meaningful change on the Functional Assessment of Cancer Therapy-Biologic Response Modifiers (FACT-BRM) instrument. Value Health. 2005 Mar-Apr;8(2):117-27. doi: 10.1111/j.1524-4733.2005.08202.x. PMID 15804320
- [Background] Webster K, Cella D, Yost K. The Functional Assessment of Chronic Illness Therapy (FACIT) Measurement System: properties, applications, and interpretation. Health Qual Life Outcomes. 2003 Dec 16;1:79. doi: 10.1186/1477-7525-1-79. PMID 14678568
- [Background] Cella D, Li JZ, Cappelleri JC, Bushmakin A, Charbonneau C, Kim ST, Chen I, Motzer RJ. Quality of life in patients with metastatic renal cell carcinoma treated with sunitinib or interferon alfa: results from a phase III randomized trial. J Clin Oncol. 2008 Aug 1;26(22):3763-9. doi: 10.1200/JCO.2007.13.5145. PMID 18669464
- [Background] Fairclough DL, Cella DF. Functional Assessment of Cancer Therapy (FACT-G): non-response to individual questions. Qual Life Res. 1996 Jun;5(3):321-9. doi: 10.1007/BF00433916. PMID 8763800
- [Background] Jaeschke R, Singer J, Guyatt GH. Measurement of health status. Ascertaining the minimal clinically important difference. Control Clin Trials. 1989 Dec;10(4):407-15. doi: 10.1016/0197-2456(89)90005-6. PMID 2691207
- [Background] Guyatt GH, Osoba D, Wu AW, Wyrwich KW, Norman GR; Clinical Significance Consensus Meeting Group. Methods to explain the clinical significance of health status measures. Mayo Clin Proc. 2002 Apr;77(4):371-83. doi: 10.4065/77.4.371. PMID 11936935
- [Background] Cella D, Hahn EA, Dineen K. Meaningful change in cancer-specific quality of life scores: differences between improvement and worsening. Qual Life Res. 2002 May;11(3):207-21. doi: 10.1023/a:1015276414526. PMID 12074259
- [Background] Brucker PS, Yost K, Cashy J, Webster K, Cella D. General population and cancer patient norms for the Functional Assessment of Cancer Therapy-General (FACT-G). Eval Health Prof. 2005 Jun;28(2):192-211. doi: 10.1177/0163278705275341. PMID 15851773
- [Background] Rege RV. Adverse effects of biliary obstruction: implications for treatment of patients with obstructive jaundice. AJR Am J Roentgenol. 1995 Feb;164(2):287-93. doi: 10.2214/ajr.164.2.7839957.
- [Background] Kramer HJ. Impaired renal function in obstructive jaundice: roles of the thromboxane and endothelin systems. Nephron. 1997;77(1):1-12. doi: 10.1159/000190241. PMID 9380222
- [Background] Jiang WG, Puntis MC. Immune dysfunction in patients with obstructive jaundice, mediators and implications for treatments. HPB Surg. 1997;10(3):129-42. doi: 10.1155/1997/49076. PMID 9174857
- [Background] Cotton PB, Schmitt C. Quality of Life in palliative management of malignant obstructive jaundice. Scand J Gastroenterol Suppl. 1993;199:44-6. doi: 10.3109/00365529309098357. PMID 7513440
- [Background] Moss AC, Morris E, Leyden J, MacMathuna P. Malignant distal biliary obstruction: a systematic review and meta-analysis of endoscopic and surgical bypass results. Cancer Treat Rev. 2007 Apr;33(2):213-21. doi: 10.1016/j.ctrv.2006.10.006. Epub 2006 Dec 8. PMID 17157990
- [Background] Yeoh KG, Zimmerman MJ, Cunningham JT, Cotton PB. Comparative costs of metal versus plastic biliary stent strategies for malignant obstructive jaundice by decision analysis. Gastrointest Endosc. 1999 Apr;49(4 Pt 1):466-71. doi: 10.1016/s0016-5107(99)70044-1. PMID 10202060
- [Background] Fitzsimmons D, Johnson CD. Quality of life after treatment of pancreatic cancer. Langenbecks Arch Surg. 1998 Apr;383(2):145-51. doi: 10.1007/s004230050106. PMID 9641887
- [Derived] Barkay O, Mosler P, Schmitt CM, Lehman GA, Frakes JT, Johanson JF, Qaseem T, Howell DA, Sherman S. Effect of endoscopic stenting of malignant bile duct obstruction on quality of life. J Clin Gastroenterol. 2013 Jul;47(6):526-31. doi: 10.1097/MCG.0b013e318272440e. PMID 23269313